CLINICAL TRIAL: NCT01366144
Title: An Early Phase 1 Study of ABT-888 in Combination With Carboplatin and Paclitaxel in Patients With Hepatic or Renal Dysfunction and Solid Tumors
Brief Title: Veliparib, Paclitaxel, and Carboplatin in Treating Patients With Solid Tumors That Are Metastatic or Cannot Be Removed by Surgery and Liver or Kidney Dysfunction
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02500; NCI-2011-02500 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000700997; UPCI 10-115; UPCI-10-115; 8808 (Other: University of Pittsburgh Cancer Institute (UPCI)); 8808 (Other: CTEP); N01CM00100 (NIH); P30CA047904 (NIH); U01CA062490 (NIH); U01CA062502 (NIH); U01CA062505 (NIH); U01CA069856 (NIH); U01CA070095 (NIH); U01CA099168 (NIH); UM1CA186690 (NIH); UM1CA186691 (NIH); UM1CA186709 (NIH); UM1CA186716 (NIH); UM1CA186717 (NIH)
Record Dates: First submitted 2011-06-02; First posted 2011-06-03 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Breast Carcinoma; Carcinoma of Unknown Primary; Endometrial Carcinoma; Esophageal Carcinoma; Liver Failure; Lung Carcinoma; Malignant Head and Neck Neoplasm; Malignant Testicular Neoplasm; Melanoma; Metastatic Malignant Solid Neoplasm; Ovarian Carcinoma; Renal Failure; Unresectable Malignant Neoplasm; Urothelial Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Neoplasms, Unknown Primary; Endometrial Neoplasms; Esophageal Neoplasms; Liver Failure; Lung Neoplasms; Head and Neck Neoplasms; Testicular Neoplasms; Melanoma; Neoplasm Metastasis; Ovarian Neoplasms; Renal Insufficiency; Carcinoma, Transitional Cell | interventions — Carboplatin; Paclitaxel; Taxes; veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (veliparib, paclitaxel, carboplatin) (Experimental): Patients receive veliparib* PO BID on days 1-7 and paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 3. Courses repeat every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  NOTE: * All patients receive a single dose of veliparib PO on day -6 before course 1 (except patients with very severe renal dysfunction who receive veliparib on day -5 or -6 to coincide with a dialysis day).
  Interventions: Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Pharmacological Study; Drug: Veliparib

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Other: Pharmacological Study — Correlative studies
Drug: Veliparib — Given PO
  Other Names: ABT 888; ABT-888; ABT888; PARP-1 inhibitor ABT-888

SUMMARY:
This phase I trial studies the side effects and the best dose of veliparib when given together with paclitaxel and carboplatin in treating patients with solid tumors that are metastatic or cannot be removed by surgery and liver or kidney dysfunction. Veliparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving veliparib together with paclitaxel and carboplatin may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the pharmacokinetics and pharmacodynamics of ABT-888 (veliparib) in patients with varying degrees of renal or hepatic dysfunction.

II. To determine the maximum tolerated dose (MTD) of ABT-888 in combination with carboplatin and paclitaxel for patients with varying degrees of liver or kidney dysfunction.

III. To provide dosing recommendations for ABT-888 in combination with carboplatin and paclitaxel based on degree of hepatic and renal impairment.

SECONDARY OBJECTIVES:

I. To define the dose-limiting toxicity (DLT) and other toxicities associated with the use of this combination in patients with varying degrees of renal or hepatic dysfunction.

II. To evaluate the pharmacokinetic parameters of ABT-888, carboplatin, and paclitaxel when administered as a combination in patients with varying degrees of renal or hepatic dysfunction.

III. To evaluate the pharmacodynamic measurement of poly-ADP-ribosylated (PAR) and platinum adducts in tumor cells associated with the use of this combination in patients with varying degrees of renal or hepatic dysfunction.

OUTLINE: This is a dose-escalation study of veliparib.

Patients receive veliparib* orally (PO) twice daily (BID) on days 1-7 and paclitaxel intravenously (IV) over 3 hours and carboplatin IV over 30 minutes on day 3. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.

NOTE: * All patients receive a single dose of veliparib PO on day -6 before course 1 (except patients with very severe renal dysfunction who receive veliparib on day -5 or -6 to coincide with a dialysis day).

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed malignancy that is radiologically evaluable and metastatic or unresectable, for which standard curative or palliative measures do not exist or are no longer effective, and for which there is expectation of response to the combination of carboplatin/paclitaxel (i.e., lung, ovarian, breast, melanoma, head and neck, endometrial, urothelial, testicular, esophageal, carcinoma of unknown primary); for indications not listed, eligibility based on disease must be verified by the principal investigator before they are considered
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 12 weeks
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 8.0 g/dL
* Patients with all degrees of renal dysfunction are allowed including patients on hemodialysis; patients with mild to severe hepatic dysfunction are allowed as defined below:
* Total bilirubin =< 5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 10 x ULN
* For patients with a recently placed biliary stent, patients should have consistent results within a hepatic group from two laboratory readings within 3 days apart, taken at least 10 days following biliary stent placement; for patients with a biliary stent placed over 2 months ago, no obstruction or blockage can have occurred within the last 2 months
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those whose adverse event due to agents administered more than 4 weeks earlier have not resolved or stabilized; patients who have been administered ABT-888 as part of a single or combination, phase 0 or I study, should not necessarily be excluded from participating in this study solely because of receiving prior ABT-888
* Patients may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ABT-888 or other agents used in study
* Peripheral neuropathy of severity greater than grade 1
* Inability to take oral medications on a continuous basis
* Evidence of bleeding diathesis
* Patients with central nervous system (CNS) metastases must be stable after therapy for CNS metastases (such as surgery, radiotherapy or stereotactic radiosurgery) for at least 3 months and must be off steroid treatment prior to study enrollment
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with ABT-888; these potential risks may also apply to other agents used in this study
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible; however, HIV-positive patients without an acquired immune deficiency syndrome (AIDS)-defining diagnosis who are not receiving agents with the potential for pharmacokinetic (PK) interactions with ABT-888 may be eligible
* Patients with both hepatic and renal dysfunction will also be excluded
* Patients who received and progressed on the combination of carboplatin/paclitaxel will not be eligible
* Active seizure or history of seizure disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2011-06-20 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2026-03-17 (Estimated)

PRIMARY OUTCOMES:
PK parameters of veliparib | Day -6 and 3 of course 1 after veliparib dosing
  Standard quantitative and graphical statistical summaries of the derived PK parameters (e.g. area under curve and clearance) will be produced for each organ function cohort. The effect of dysfunction on pharmacokinetics will be explored by comparing each pharmacokinetic parameter across all cohorts using one-way analysis (analysis of variance) or Kruskal-Wallis test. The level of each protein will be compared between responders and non-responders using the Wilcoxon signed rank test.
MTD of veliparib in combination with carboplatin and paclitaxel, determined according to incidence of DLT as graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version (v) 4.0 | 21 days

SECONDARY OUTCOMES:
Incidence of toxicities as assessed by NCI CTCAE v4.0 | Up to 4 weeks after completion of study treatment
  The maximum grade of toxicity for each category of interest will be recorded for each patient and the summary results will be tabulated by category, grade and dose level. Severe and life-threatening toxicities and adverse event-related deaths (>= grade 3) will be described on a patient-by-patient basis and will include any relevant baseline data.
Response rate as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | Up to 4 weeks after completion of study treatment
  Responses will be tabulated by disease diagnosis and by dose level. 95% confidence limits will also be reported on the response rates.
Incidence of stable disease as assessed by RECIST version 1.1 | Up to 4 weeks after completion of study treatment
  Incidence of stable disease will be tabulated by disease diagnosis and by dose level.
Time to progression | Up to 4 weeks after completion of study treatment
  Displayed for all patients and for patients who have responded; no formal statistical analysis is planned.

OTHER OUTCOMES:
Change in PAR levels | Baseline to up to 4 weeks
  Descriptive statistics (mean, standard deviation, median, range) for measurements of PAR levels will provided with 95% confidence intervals (CIs). When sample size permits, a formal statistical test using the Wilcoxon signed rank test will be used to compare the post treatment PAR levels to the baseline levels. When feasible, the level will be compared between responders and non-responders using the Wilcoxon signed rank test.
Change in gamma-H2AX levels | Baseline to up to 4 weeks
  Descriptive statistics (mean, standard deviation, median, range) for measurements of gamma-H2AX levels will provided with 95% CIs. When sample size permits, a formal statistical test using the Wilcoxon signed rank test will be used to compare the post treatment PAR levels to the baseline levels. When feasible, the level will be compared between responders and non-responders using the Wilcoxon signed rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Hussein A Tawbi, Principal Investigator — University of Pittsburgh Cancer Institute (UPCI)
Locations (17):
- United States (17):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - City of Hope South Pasadena, South Pasadena, California
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Case Western Reserve University, Cleveland, Ohio
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin